CLINICAL TRIAL: NCT02026167
Title: SCI-CARE (Northwest Regional Spinal Cord Injury Site Specific Project)
Brief Title: Spinal Cord Injury Collaborative Care Study
Acronym: SCI-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Bombardier, Professor, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001791
Record Dates: First submitted 2013-12-26; First posted 2014-01-01 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Spinal Cord Injury
Keywords: Chronic Pain; Mood; Physical Activity
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): No intervention, usual care
- Intervention (Experimental): Collaborative care with Health Care Assistant
  Interventions: Behavioral: Collaborative Care

INTERVENTIONS:
Behavioral: Collaborative Care — Addition of a Health Care Assistant to treatment team, case review by expert panel of supervisors, non-medical interventions
  Arms: Intervention

SUMMARY:
The objective of this study is to test the effectiveness of a collaborative care approach to improving outpatient treatment for inactivity, chronic pain and depression as a way of improving overall Quality of Life for patients with SCI.

DETAILED DESCRIPTION:
Individuals with SCI were treated by a care manager who worked in collaboration with the participant's physician to decrease pain, decrease depression symptoms, and/or to increase physical activity. This was done by collaborating on current treatments to make sure that they are being as effective as possible and by providing non-pharmacological treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* diagnosis of traumatic spinal cord injury by medical record review
* receives primary SCI care from a provider at the University of Washington or Harborview Medical Center's Rehabilitation Outpatient Clinic
* positive screening for pain related to SCI diagnosis and/or
* positive screening for low mood and/or
* negative screening for physical activity levels
* able to speak and understand English

Exclusion Criteria:

* psychiatric condition that would interfere with participation
* major surgery in the next 8 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline, 4 months
  Quality of Life is assessed via telephone interviews at baseline and 4 months.

SECONDARY OUTCOMES:
Change in Pain | Baseline, 4 months, 8 months
  Pain is assessed via telephone interview at baseline, 4 months, and 8 months.
Change in Mood | Baseline, 4 months, 8 months.
  Mood assessed via telephone interviews at baseline, 4 months, and 8 months.
Change in Physical Activity | Baseline, 4 months, 8 months
  Physical activity is assess via telephone interview at baseline, 4 months, and 8 months.
Change in Quality of Life | Baseline, 8 months
  Change in QOL from baseline to 8 months will be compared between groups
Adverse events | baseline to 4 months
  The number of cases with serious or non-serious adverse events in the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Bombardier, Ph.D., Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: General study information on the Northwest Regional SCI System website — http://sci.washington.edu/scicare/